CLINICAL TRIAL: NCT00576355
Title: Adjunctive Psychotherapy for Teens With Bipolar Disorder
Brief Title: Interpersonal and Social Rhythm Therapy for Adolescents With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH070570 (NIH); K23MH070570 (NIH); 5K23MH070570-03 (NIH); DDTR BK-TKAR
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Bipolar Disorder
Keywords: Adolescent; Psychopathology; Interpersonal Therapy; Interpersonal and Social Rhythm Therapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment As Usual (TAU)
- 1 (Experimental): Participants will receive interpersonal and social rhythm therapy for adolescents
  Interventions: Behavioral: Interpersonal and Social Rhythm Therapy for Adolescents (IPSRT-A)

INTERVENTIONS:
Behavioral: Interpersonal and Social Rhythm Therapy for Adolescents (IPSRT-A) — IPSRT-A involves 20 weeks of individual therapy, incorporating informed psychological, behavioral, and practical strategies adapted to the developmental needs of adolescents.
  Arms: 1
Behavioral: Treatment As Usual (TAU) — TAU includes the offering of educational information about bipolar disorder and referral to a mental health provider.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of interpersonal and social rhythm therapy in treating adolescents with a bipolar spectrum disorder

DETAILED DESCRIPTION:
Bipolar disorder is a brain disorder that causes dramatic changes in a person's mood and energy. Bipolar spectrum disorders, including bipolar I, II, and not-otherwise-specified (NOS) disorders, usually form in late adolescence or early adulthood and require treatment for the rest of a person's life. People with a bipolar spectrum disorder undergo periods of extreme happiness and extreme sadness, known as episodes of mania and depression. Psychotherapy has proven an effective adjunct treatment to medications for people with bipolar disorder. Interpersonal and social rhythm therapy (IPSRT) is a specific type of psychotherapy that focuses on improving problems in interpersonal relationships that are related to a person's symptoms. Researchers believe that IPSRT helps people have more regular patterns of sleep, eating, and other activities that act to set a person's biological clock. This study will specifically adapt IPSRT to the developmental needs of adolescents and will determine the effectiveness of this approach in treating adolescents with a bipolar spectrum disorder.

Participants in this study will be randomly assigned to receive interpersonal and social rhythm therapy for adolescents (IPSRT-A) or treatment as usual (TAU). Participants assigned to IPSRT-A will take part in 18 sessions of IPSRT over a 20-week period. Beginning with the first session, participants will meet with a therapist weekly for 16 weeks and then every other week for 4 weeks. Each IPSRT session will last about 45 to 60 minutes, and parents will be asked to accompany the child to 2 to 4 of these sessions. During IPSRT sessions, the therapist will talk with participants about their relationships and how they relate to symptoms; work with participants to help improve understanding of how their social and sleep routines relate to symptoms; and teach participants about bipolar disorder. Participants assigned to TAU will be given educational information about bipolar disorder and its treatment. They will then be referred to a mental health provider for usual care treatment.

All participants and parents will complete questionnaires about symptoms every 4 weeks during the study. Follow-up assessments will occur at the end of treatment and again at Months 3 and 6 post-treatment. These assessments will last between 60 and 90 minutes and will include completing an interview and questionnaires. Participants will also be asked for permission to obtain grade point average (GPA) and attendance records from their schools.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of bipolar spectrum disorder: type I, type II, or NOS
* Currently meets DSM-IV criteria for a depressed, manic, hypomanic, or mixed episode
* Youth assent/parental consent to outpatient psychotherapy for treatment of bipolar disorder
* Adequate access to transportation or close proximity in order to participate in therapy

Exclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizophreniform, or schizoaffective disorders
* Developmentally delayed
* Actively psychotic, suicidal, homicidal, or engages in repeated parasuicidal behaviors
* History of chronic suicidality (e.g., more than three suicidal gestures in the year prior to study entry)
* Neurological or other medical disorder that could potentially cause or complicate presenting psychiatric symptoms
* Meets current DSM-IV criteria for drug or alcohol abuse or dependence
* Life circumstances that would prohibit ability to participate, including absence of shelter or impending jail/prison for more than 2 weeks during study
* Parent/legal guardian refusal to participate with the adolescent

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale for Children | Measured at pretreatment, every 4 weeks during treatment, post-treatment, and 3 and 6 month follow-ups

SECONDARY OUTCOMES:
Mania Rating Scale (MRS), Beck Depression Inventory (BDI),Child Behavior Checklist (CBCL), Youth Self-Report Form (YSR), Social Adjustment Scale for Adolescents (SAS-SR-A), Conflict Behavior Questionnaire (CBQ) | Measured at pretreatment, post-treatment, 6 month follow-up, and various other times throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hlastala, PhD, Principal Investigator — University of Washington, Children's Hospital and Regional Medical Center
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States